CLINICAL TRIAL: NCT00663195
Title: Effects of Spironolactone on Circulating MMPs in Patients With Chronic Heart Failure
Brief Title: Effects of Spironolactone on Matrix Metalloproteinases (MMPs) in Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tottori University Hospital (Other)
Responsible Party: Kazuhide Ogino, Center for Clinical Residency Program, Tottori University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: #344
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Chronic Stable Heart Failure
Keywords: heart failure; fibrosis; MMP; spironolactone; furosemide
MeSH Terms: conditions — Heart Failure; Fibrosis | interventions — Spironolactone; Furosemide

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: spironolactone + furosemide — spironolactone 25mg/day, 16 weeks and furosemide 20mg/day, 16 weeks

SUMMARY:
The purpose of this study is to evaluate the effects of spironolactone on circulating MMP levels and insulin resistance in patients with chronic heart failure.

DETAILED DESCRIPTION:
Myocardial fibrosis is observed in failing hearts. MMPs are considered markers of fibrosis. Recently, circulating MMPs can be measured and are elevated in patients with chronic heart failure (CHF). It has been reported that spironolactone improves myocardial fibrosis in CHF animal models. Therefore, the purpose of this study is to evaluate the effects of spironolactone on circulating MMP levels in patients with chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* chronic stable heart failure

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-01; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
MMP levels | 16 weeks